CLINICAL TRIAL: NCT04699370
Title: The Added Value of Cognition-targeted Exercise Versus Symptom-targeted Exercise for Multiple Sclerosis Fatigue: Randomized Controlled Trial
Brief Title: The Added Value of Cognition-targeted Exercise Versus Symptom-targeted Exercise for Multiple Sclerosis Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ibrahim Moustafa, Associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cairo 2021
Record Dates: First submitted 2021-01-02; First posted 2021-01-07 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Physical and Rehabilitation Medicine
Keywords: Randomized controlled trial; Multiple Sclerosis; Fatigue; Cognitive Behavioral Therapy; exercise
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Motor Activity | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: A prospective, parallel-group, randomized clinical trial participants will be randomly assigned to the control group or intervention group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cognition-targeted exercise (Experimental): The patients in this group will receive cognitive behavior therapy in addition to cognition-targeted exercise .
  Cognitive behavior therapy will be designed on the basis of van Kessel's model . The main objective of this treatment will be challenging all external factors (e.g. behavioral, cognitive, and affective factors) envisioned to play a role in the development and persistence of fatigue in MS patients. The treatment sessions will be directed individually.
  For Cognition- targeted exercise , all standardized physical therapy exercises will be performed in a time-contingent rather than in a symptom-contingent way .
  Interventions: Other: cognition-targeted exercise; Behavioral: Cognitive behavioral therapy
- symptom-targeted exercise (Active Comparator): The patients in this group will receive cognitive behavior therapy in addition to symptom-targeted exercise .
  Cognitive behavior therapy will be designed on the basis of van Kessel's model . The main objective of this treatment will be challenging all external factors (e.g. behavioral, cognitive, and affective factors) envisioned to play a role in the development and persistence of fatigue in MS patients. The treatment sessions will be directed individually.
  For symptom- targeted exercise, All Standardized physical therapy exercises will be performed in a symptom-contingent way ("Stop or adjust the exercise when it hurts").
  Interventions: Behavioral: Cognitive behavioral therapy; Other: Standardized physical therapy

INTERVENTIONS:
Other: cognition-targeted exercise — All Standardized physical therapy exercises will be performed in a time-contingent .
  Goal setting is essentially done together with the patient, focussing on functionality instead of fatigue relief. Progression to a next level of (more difficult) exercises will be preceded by an intermediate phase of motor imagery.
  The treating physical therapist will be advised to address patients' cognitions about their problems during the cognition-targeted exercise training, so that patients will have positive perceptions regarding their illness and treatment outcome.
  The treating physical therapist will be advised to discuss the patient's perceptions about each exercise. This include discussion of the anticipated consequences of the exercises and challenging the patient's cognitions in relation to the exercises
  Arms: cognition-targeted exercise
Behavioral: Cognitive behavioral therapy — In the first and second sessions, patients will learn about fatigue-related symptoms as well as Cognitive behavioral therapy and its effectiveness. The third and fourth sessions will be devoted on the introduction of behavioral strategies. The fifth session will introduce cognitive strategies to decrease fatigue. The last three sessions will be about how to adopt the proposed strategies consistently.
Other: Standardized physical therapy — The standardized physical therapy will consist of eight half-hour individualized face to face physiotherapy sessions, over a 4-week period. this program will consist of twice-weekly supervised general aerobic, strengthening and flexibility exercise sessions .This exercise program is reflective of the general exercises typically undertaken within routine clinical practice.
  Arms: symptom-targeted exercise

SUMMARY:
Introduction: Multiple sclerosis (MS) has a wide range of physiological and neuropsychological symptoms. Over 75% of MS patients complain about fatigue, which for many is one of their most debilitating symptoms, having a substantial impact on their quality of life and ability to carry out day-to-day tasks. Previous investigations on the effectiveness of different types of psychotherapy on MS fatigue are extremely limited. The aim of this study was to investigate the added value of cognition-targeted exercise versus symptom-targeted exercise for Multiple Sclerosis fatigue

DETAILED DESCRIPTION:
Patients with fatigue symptoms (score of ≥5 on Fatigue Scale) will be randomly assigned into experimental (n=30) and control (n=30) groups. The subjects in the experimental group will receive eight 50-minute sessions of weekly cognitive behavior therapy based on van Kessel's model in addition cognition-targeted exercise program , whereas the patients in the control group will receive eight 50-minute sessions of weekly CBT in addition to standardized physiotherapy program . A standardized program of physiotherapy exercises will consist of twice-weekly supervised general aerobic, strengthening and flexibility exercise sessions. This exercise program is reflective of the general exercises typically undertaken within routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis by a neurologist which incorporate clinical features with magnetic resonance scanning.
* Being within normal or average dysfunction and excluding those scoring ≤6 in the Expanded Disability Status Scale (EDSS);
* Being identified as a case level of fatigue; fatigue score of 4 or greater on the Fatigue Scale (FS);

Exclusion Criteria:

* Patients with any serious psychological disorders (including psychotic disorders or active substance abuse), or those with any chronic illness that may be contributing to fatigue were excluded.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Change in Modified Fatigue Impact Scale | pre-treatment , at 4-week,and after three months
  The Modified Fatigue Impact Scale is a modified form of the Fatigue Impact Scale based on items derived from interviews with MS patients concerning how fatigue impacts their lives. Items on the Modified Fatigue Impact Scale are aggregated into three subscales (physical, cognitive, and psychosocial), as well as into a total Modified Fatigue Impact Scale score. All items are scaled so that higher scores indicate a greater impact of fatigue on a person's activities.

SECONDARY OUTCOMES:
Change in Work and Social Adjustment Scale | pre-treatment , at 4-week,and after three months
  The Work and Social Adjustment Scale , which assessed fatigue-related impairment in relation to a number of areas of the person's life. The maximum score is 40 .lower score is better
Change in Hospital Anxiety and Depression Scale | pre-treatment , at 4-week,and after three months
  The Hospital Anxiety and Depression Scale , a commonly used self-report instrument for detecting states of depression and anxiety in patients with medical illnesses. scores of less than 7 indicate non-cases and high scores indicate more anxiety and depression
Change in Perceived Stress Scale | pre-treatment , at 4-week,and after three months
  the Perceived Stress Scale will be included to assess whether the degree to which patients appraised situations in their lives as stressful changed after the intervention. Individual scores on the Perceived Stress Scale can range from 0 to 40 with higher scores indicating higher perceived stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
no plan to make individual participant data (IPD) available to other researchers